CLINICAL TRIAL: NCT02925312
Title: MedStar Pathway to Diabetes Control Demonstration Project: Type 2 Diabetes Boot Camp
Brief Title: MedStar Health Type 2 Diabetes Pathway to Control
Acronym: T2DMBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Michelle Magee, Director, MedStar Diabetes Institute, Medstar Health Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-191
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Results first posted 2020-07-17 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes Mellitus; Hyperglycemia
Keywords: Diabetes Care Management; Chronic Care Model; Resources Utilization; Hemoglobin A1C; Hospitalizations; Emergency Room Visits; Cost analysis; Return on Investment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Patients receive the full diabetes pathway intervention consisting of: individualized diabetes self-management education and support; T2DM meds management by clinician-supervised diabetes educators using an evidence-based algorithm and FDA approved anti-hyperglycemic agents; near, real-time blood glucose monitoring, delivered via a combination of two in-person and weekly remote (telephone/text) visits.
  Interventions: Other: Diabetes Pathway
- Matched controls (No Intervention): Patients receive standard of care from their primary care provider. Usual care visits are typically conducted quarterly per national guidelines for management of T2DM in adults, or more frequently as needed.

INTERVENTIONS:
Other: Diabetes Pathway — Medication algorithm, survival skills education, enhanced patient-provider communication facilitated by near, real-time blood glucose monitoring
  Other Names: Diabetes Boot Camp
  Arms: Intervention

SUMMARY:
A Diabetes Institute (MDI), in partnership with key stakeholders-including Primary Care Providers- in a northeastern US regional, mixed-payer healthcare system), seeks to implement an evidence-based, technology-enabled, innovative, and integrated diabetes care management pathway (Boot Camp) for adult patients with uncontrolled type 2 diabetes (A1C>/=9%) which will demonstrate improvement in diabetes clinical and health resources utilization outcomes.

DETAILED DESCRIPTION:
* The program is designed to integrate type 2 diabetes specialty services into Primary Care practices to support PCPs and their patients in improving a spectrum of diabetes-related outcomes.
* High-risk patients from Primary Care practices who have uncontrolled type 2 diabetes and meet the target population inclusion and exclusion criteria will be invited to participate in an intensive and concise "BOOT CAMP" medication management and education intervention of ~4-8 weeks duration.
* The intervention will consist of three key components: (1) intensive, algorithm-based medication management (Appendix A), based on continuous review and management of blood sugars; (2) survival skills diabetes self-management education based on knowledge deficits identified on the KNOW Diabetes knowledge survey; (3) enhanced patient-provider communication, all provided by Endocrinologist supervised allied health professionals (in this instance CDEs).
* Survival skills DSME will focus on nutrition and meal plan basics, blood glucose targets, taking medications as prescribed, hyper- and hypoglycemia recognition and treatment, and when to seek medical help.
* The intervention is initiated with one to two face-to-face meetings with the CDE, at which the patient's readiness to change is assessed.
* These are followed by virtual meetings though a variety of media based on patient preference and health literacy (largely telephone and text messaging).
* Various technology tools are used to facilitate patient engagement, access and attainment of glycemic targets, including smart meters, virtual meeting platforms, web-based education content and surveys administration via tablets, etc.
* Near real-time transmission of blood glucose data using a cellular-enabled blood glucose monitoring system sends all glucose results to a web-based dashboard accessed daily by the Boot Camp educators.
* Concurrent matched charts of patients receiving standard care at the three MedStar locations will serve as a basis of comparison in assessing the impact of MDI on clinical and education outcomes and process of care.
* Based on patient progress towards improved glycemic control, the patient will 'graduate' from the program and the CDE will refer the patient back to their PCP in 8-12 weeks with a full report of medication changes, blood glucose readings and further diabetes management recommendations eg referrals; further DSME, etc.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes for >=1 year
* Active practice patient
* A1C > 9.0% at their last visit to Medical Home, ED or hospital admission plus one more high risk factor (ED visit or hospitalization in past 12 mos)
* Primary Care Provider willing to have patient enter the program
* Patient is able and willing to participate in the program and exhibits readiness to change DM self-management
* Proficient in English

Exclusion Criteria:

* Known history of DKA
* No MedStar PCP visit within past 12 months
* Endocrine or Diabetes Education consult referral order in the past 6 months which resulted in Endo visit(s) or DSME visit(s) documented in chart or self-reported by patient during initial screen
* Active additional medical issues which in the opinion of the care team would preclude concentrating on BG control and/or would predispose to ED visits and/or hospital admits independent of glycemic control, e.g.: severe CHF, severe COPD; severe mental illness.
* Resident of skilled nursing facility, nursing home or receiving home health care services.
* Active cancer in the preceding 3 years excluding nonmalignant basal cell cancer
* Supraphysiologic doses of glucocorticoids (hydrocortisone > 30mg/day; prednisone > 5-6mg daily; dexamethasone > 2mg daily).
* Pregnant or anticipates attempting conception in the following year
* Patient and/or custodial caregiver unwilling and/or unable to participate in program-related activities

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06-30 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle F Magee, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request to the PI including provision of details of how the IPD will be utilized by the requestor, the study team will decide whether to release the IPD. The study protocol, SAP, ICF and clinical study report will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon final completion of reporting of main study results the study protocol, SAF, ICF and CSR will be available for 5 years.
Access Criteria: Deidentified data for scientific use that may contribute to the body of evidence to inform diabetes care management.

REFERENCES:
- [Background] Magee MF, Baker KM, Fernandez SJ, Huang CC, Mete M, Montero AR, Nassar CM, Sack PA, Smith K, Youssef GA, Evans SR. Redesigning ambulatory care management for uncontrolled type 2 diabetes: a prospective cohort study of the impact of a Boot Camp model on outcomes. BMJ Open Diabetes Res Care. 2019 Nov 13;7(1):e000731. doi: 10.1136/bmjdrc-2019-000731. eCollection 2019. PMID 31798894
- [Derived] Montero AR, Toro-Tobon D, Gann K, Nassar CM, Youssef GA, Magee MF. Implications of remote monitoring Technology in Optimizing Traditional Self-Monitoring of blood glucose in adults with T2DM in primary care. BMC Endocr Disord. 2021 Nov 10;21(1):222. doi: 10.1186/s12902-021-00884-6. PMID 34758807

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Patients receive the full diabetes pathway intervention
  Diabetes Pathway: Medication algorithm, survival skills education, enhanced patient-provider communication
- Matched Controls: patients receive standard of care
Period: Overall Study
Arm/Group | Intervention | Matched Controls
Started | 125 | 294
Completed | 98 | 294
Not Completed | 27 | 0
Not completed — Lost to Follow-up | 25 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Matched Controls | Total
Number analyzed (Participants) | 121 | 294 | 415
Age, Customized [Count of Participants; unit: Participants]
  age between 21 and 75 | 121 | 294 | 415
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 162 | 229
  Male | 54 | 132 | 186

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Hemoglobin A1C From Baseline to 3 Months
Description: Comparison of the percentage change in A1C from baseline to 3 months between the intervention and the control group
Time Frame: 3 months
Population: Boot camp completers during the study period were compared to concurrent, propensity-matched chart controls.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Intervention | Matched Controls
Number analyzed (Participants) | 121 | 294
percentage | 3.08 (2.01) | 1.64 (1.97)
Statistical Analysis 1: Comparison: Intervention vs Matched Controls; The study was powered to detect a difference of 0.5 in the change in HbA1c with SD=2 with 80% power at alpha=0.05 with a sample size of 128 in each group (paired t-test). Differences in patient characteristics and the unadjusted differences in the outcome measures between the intervention and control groups were tested using linear mixed models, McNemar tests and conditional logistic models due to matching; Test type: Superiority; p = 0.05, McNemar

2. Secondary Outcome: Risk of Experiencing a Composite Endpoint of All Cause ED Visits and Hospitalizations at 6 Months Post Intervention vs 6 Months Pre-intervention for Cases and Controls.
Description: Health care utilization measure. We compared the risk of experiencing an emergency room and/or hospital visit at 6 months from baseline for both groups. this was done by calculating he Incidence Risk Ratio of ED visits/hospitalizations for intervention and control patients to assess whether the pathway impacted the risk for ED visits/hospitalizations at 6 months from baseline and comparing them. We looked at these measures for the 6-month period that preceded the baseline visit and the 6-month period that followed the baseline visit.
Time Frame: 6 months
Population: Poisson Regression Models of all utilizations (ED + hospitalization) at 6-month visits by Study Groups: Incidence rate ratios (IRRs) reported. In the six months after enrollment, controls are expected to have 0.646 admissions on average, and cases are expected to have 56.8% of the number of admissions that the controls had, or a reduction of 43.2%
Measure: Number (95% Confidence Interval); unit: ratio of risk incidences
Arm/Group | Intervention | Matched Controls
Number analyzed (Participants) | 98 | 294
ratio of risk incidences | 0.568 [0.398 to 0.812] | 0.646 [0.561 to 0.745]

3. Secondary Outcome: Adherence to Prescribed Diabetes Medications
Description: Change in Adherence to Diabetes Medications as Measured Using MMS From Baseline to 3 Months for Intervention Subjects
Time Frame: 90 days
Population: This outcome measure was eliminated during the course of the study and data was not collected
Arm/Group | Intervention | Matched Controls
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Frequency of Eye Exams
Description: Change in the Proportion of Patients Receiving an Eye Exam in the 6 Months Following the Start of the Intervention as Compared to Baseline and to Concurrent Chart Controls
Time Frame: 90 days
Population: Technology to perform eye exams in primary care offices was not deployed as had been anticipated, therefore data was not collected for this outcome
Arm/Group | Intervention | Matched Controls
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Intervention | Matched Controls
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/294
Other Adverse Events (participants affected / at risk) | 0/121 | 0/294

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes